CLINICAL TRIAL: NCT06398912
Title: Studying Newborns' Brain Activity in the NICU Through a Musical Intervention: the Role of Fundamental Frequency
Acronym: FunFreqNICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athens General Children's Hospital "Pan. & Aglaia Kyriakou" (Other)
Responsible Party: Principal Investigator, Dr Angeliki Nika, Neonatologist - Director of NICU, Athens General Children's Hospital "Pan. & Aglaia Kyriakou"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09th/04-05-2023 (Θ: 9)
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Premature Birth
Keywords: Premature Infants; Music; Brain Development; Pediatrics; Neonatology
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention (Experimental): Participants will be exposed to an organized sound stimulus (music) during the EEG measurement
  Interventions: Other: Music Based Intervention
- Control Group (No Intervention): Participants will not be exposed to an organized sound stimulus at any point of the EEG measurement

INTERVENTIONS:
Other: Music Based Intervention — Measuring how the fundamental frequency of differential music facilitators (mother, father, male and female music therapist) impacts the premature infant brain
  Other Names: Fundamental Frequency and Brain Development Intervention
  Arms: Music Intervention

SUMMARY:
This research project stands to the intersection of neonatology, neuroscience, and music based interventions (MBIs), exploring the impact of structured sound on the brain activity of premature newborns in Neonatal Intensive Care Units (NICU). It embarks on a pioneering investigation to decipher how variations in musical stimuli, particularly those that differ in human profiles (gender and kinship) and fundamental frequencies, affect the short-term electroencephalographic (EEG) footprint of these vulnerable infants. The project aims to uncover profound insights into the therapeutic potential of music within neonatal care, thereby advancing our understanding of neurodevelopmental interventions for premature infants.

DETAILED DESCRIPTION:
Research Design and Methodology

Adopting an exploratory/randomized control trial (RCT) design, this study is meticulously planned to evaluate the effects of musical interventions on premature infants housed within a NICU setting. Therefore, participants, specifically newborns born at ≤ 32 weeks of gestation who meet stringent inclusion criteria, are randomly assigned to either an intervention group that receives structured musical interventions for a week or a control group that does not receive any musical stimulation. This methodological approach ensures a controlled examination of the intervention's efficacy, attributing observed neurophysiological changes directly to the musical stimuli.

Data Collection Protocol

The data collection protocol employs a dual approach: quantitative EEG for capturing the infants' brain activity and qualitative video recordings to document the dynamic interactions between the infants and the music facilitators. This multifaceted strategy ensures a comprehensive analysis of the effects of musical interventions, facilitated by a diverse group of individuals including male and female music therapists, and the infants' parents. Such diversity allows for a nuanced exploration of how different human profiles influence the intervention's impact on brain activity patterns.

Tools for Data Collection

The primary instrument for data collection is an 6-channel EEG system, chosen for its precision in measuring the complex electrical dynamics of the infants' brains. This is complemented by a high definition video camera that aims to capture the qualitative dimensions of the intervention, such as the infants' behavioral responses and the nuanced interaction dynamics between the infant and the facilitator. Together, these tools promise a holistic dataset that bridges the gap between neurophysiological and behavioral observations.

Data Analysis Protocol

The data analysis framework is comprehensive, incorporating (tentatively) a Repeated Measures Analysis of Variance (ANOVA) to scrutinize brain activity across different conditions, facilitators and qEEG features. This is to dissect the EEG data across the available condition variables, identifying specific patterns and variations indicative of the musical stimuli's impact.

Significance and Expected Outcomes

By melding advanced methodological design with innovative data collection and analysis techniques, the project is uniquely positioned to elucidate the neurodevelopmental benefits of musical interventions for premature infants in the NICU environment.

ELIGIBILITY:
Inclusion Criteria:

* Born at (equal or less than) 32 weeks of gestation
* Absence of auditory insufficiency in the 8th cranial nerve and excessive pathology in the brainstem
* Negative bilateral "transient evoked otoacoustic emissions," indicating unresponsiveness of the inner ear to an acoustic stimulus.
* Weighing 1000 grams or more
* In stable health conditions with no imminent risk of death
* Not sedated
* Absence of neonatal sepsis.
* No congenital, genetic, or chromosomal abnormalities.
* No nuclear jaundice.
* No maternal use of illicit drugs during pregnancy.
* No necessity for mechanical ventilation that creates excessive noise (i.e., high-frequency oscillatory ventilation).
* No need for sedative drug administration to the neonate.
* Absence of endocrine disorders (e.g., congenital hypothyroidism).

Exclusion Criteria:

* If a newborn is diagnosed with a disease or dysfunction during the study and the medical staff recommends their removal, they will be automatically excluded from the recruited sample.
* Use of other music stimulation during the implementation of the intervention period

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
qEEG features changes before, during and after the delivery of the musical intervention correlated to the fundamental frequency of the signing voice of the music facilitators | up to 18 months
  a predefined set of qEEG features (rEEG, coherence, spectral power etc) will be measured and analyzed via a 6 channels EEG unit in the NICU,

CONTACTS AND LOCATIONS:
Locations (1):
- Panagiotis and Aglaia Kyriakou Childrens Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Papatzikis E, Dimitropoulos K, Tataropoulou K, Kyrtsoudi M, Pasoudi E, O'Toole JM, Nika A. The father's singing voice may impact premature infants' brain more than their mother's: A NICU single-arm exploratory study protocol and preliminary data on a singing and EEG framework based on the fundamental frequency of voice and kinship. PLoS One. 2025 Aug 14;20(8):e0328211. doi: 10.1371/journal.pone.0328211. eCollection 2025. PMID 40811513